CLINICAL TRIAL: NCT02647320
Title: A Randomized, Double-Blind, Placebo-Controlled With Active Comparator, 12-Week Study of DS-8500a in Subjects With Type 2 Diabetes Mellitus on Metformin
Brief Title: 12-Week Study of DS-8500a in Subjects With Type 2 Diabetes Mellitus on Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DS8500-A-U202
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; interventional; double blind; phase 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; firuglipel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- DS-8500a 25mg (Experimental): One DS-8500a 25 mg tablet, 2 placebo tablets, and one placebo capsule in a once-daily oral dose
  Interventions: Drug: DS-8500a 25mg; Drug: Placebo Tablet; Drug: Placebo Capsule
- DS-8500a 50 mg (Experimental): Two DS-8500a 25 mg tablets, 1 placebo tablet, and one placebo capsule in a once-daily oral dose
  Interventions: Drug: DS-8500a 25mg; Drug: Placebo Tablet; Drug: Placebo Capsule
- DS-8500a 75 mg (Experimental): Three DS-8500a 25 mg tablets and one placebo capsule in a once-daily oral dose
  Interventions: Drug: DS-8500a 25mg; Drug: Placebo Capsule
- Placebo (Placebo Comparator): Three placebo tablets and one placebo capsule in a once-daily oral dose
  Interventions: Drug: Placebo Tablet; Drug: Placebo Capsule
- Sitagliptin 100 mg (Active Comparator): Three placebo tablets and one sitagliptin 100 mg over-capsule in a once-daily oral dose
  Interventions: Drug: Sitagliptin 100 mg; Drug: Placebo Tablet

INTERVENTIONS:
Drug: Sitagliptin 100 mg — Two sitagliptin 50 mg tablets, over-encapsulated to provide a once-daily dose of 100 mg, for oral administration
  Other Names: Januvia
  Arms: Sitagliptin 100 mg
Drug: DS-8500a 25mg — DS-8500a 25mg tablet for oral administration
  Other Names: Investigational product
  Arms: DS-8500a 25mg; DS-8500a 50 mg; DS-8500a 75 mg
Drug: Placebo Tablet — Placebo matching DS-8500a tablet for oral administration
  Other Names: Placebo
  Arms: DS-8500a 25mg; DS-8500a 50 mg; Placebo; Sitagliptin 100 mg
Drug: Placebo Capsule — Placebo matching sitagliptin over-capsule for oral administration
  Other Names: Placebo
  Arms: DS-8500a 25mg; DS-8500a 50 mg; DS-8500a 75 mg; Placebo

SUMMARY:
The hypothesis of this Phase 2, 12-week study, is that DS-8500a will improve glycemic control relative to placebo, based on changes in HbA1c, with acceptable safety and tolerability, in patients with Type 2 Diabetes Mellitus (T2DM) who are treated with metformin.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent and adhere to the study visit schedule and treatment
* Diagnosed with Type 2 diabetes mellitus as defined in the American Diabetes Association Standards of Medical Care in Diabetes 2015
* Male or female ≥ 18 and ≤ 70 years of age
* Screening fasting C-peptide > 0.5 ng/mL
* Women of child bearing potential (WOCBP) must be willing to use double-barrier contraception for the entire study
* WOCBP must have a negative pregnancy test (human chorionic gonadotropin, beta subunit [βhCG]) before entering the Lead-in Period
* Body mass index ≥ 25 kg/m2 and ≤ 45 kg/m2 at the Screening Visit
* On stable (≥ 8 weeks) metformin monotherapy ≥ 1000 mg/day
* Screening HbA1c ≥ 7.0% and ≤ 10%
* Taking ≥ 80% and ≤ 120% of both dispensed DS-8500a placebo tablets and sitagliptin placebo capsules during the Lead-in Period

Exclusion Criteria:

* History of type 1 diabetes and/or history of ketoacidosis
* History of insulin use for > 2 weeks within 2 months prior to the Screening Visit
* Two or more readings of fasting Self-monitoring of Blood Glucose (SMBG) > 240 mg/dL or worsening symptoms of hyperglycemia with one SMBG level of > 240 mg/dL during the second week of Lead-in Period, confirmed by laboratory measurement
* Screening hemoglobin <12 g/dL for males and <11 g/dL for females
* Blood donation within 2 months prior to the Screening Visit or plans to donate blood or blood products during the study
* Subjects after bariatric surgery or any gastric bypass
* Screening thyroid stimulating hormone (TSH) levels not within normal range (based on reference laboratory values )
* Screening Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) > 2.0 x upper limit of normal (ULN), and/or total bilirubin > 1.5 x ULN. If a subject has total bilirubin > 1.5 ULN, unconjugated and conjugated bilirubin fractions should be analyzed and only subjects documented to have Gilbert's syndrome may be enrolled
* Screening Serum creatinine ≥ 1.5 mg/dL for males and ≥ 1.4 mg/dL for females, or creatinine clearance (CrCl) < 50 mL/min for both males and females
* Screening Creatine kinase (CK) > 3.0 × ULN
* History of unstable angina, myocardial infarction, cerebrovascular accident, transient ischemic attack, peripheral arterial event or any revascularization procedure during the 6 months prior to the Screening Visit or planned vascular procedures or surgery during study period
* History of congestive heart failure (CHF)
* Exclusionary concomitant medications:

  a. Eight weeks prior to screening and throughout the duration of the study:
* Any diabetes medication other than metformin; any prescription or over the counter medication for weight-loss.
* Systemic corticosteroids (including nasal and inhaled), with the exception of use of topical and ophthalmic corticosteroids.
* Rosuvastatin > 20 mg daily. b. During treatment periods, additional medications will be prohibited based on potential drug-drug interaction (DDI) (see Section 5.6)
* Subjects with anticipated interruption in metformin or study drug use during the course of the clinical trial (e.g., due to an imaging procedure involving iodinated contrast media)
* Subjects in whom treatment with sitagliptin 100 mg is contraindicated ( e.g., known hypersensitivity or intolerance to sitagliptin) or may not be medically advisable (e.g., history of pancreatitis)
* Abuse of or dependence on prescription medications, illicit drugs, or alcohol within the last 1 year
* Any history of a malignancy other than basal cell carcinoma within the past 5 years
* Pregnancy or breast-feeding, or intent to become pregnant during the study period
* Known (or evidence of) infection with human immunodeficiency virus
* Any condition, laboratory abnormality, or concomitant therapy which, in the opinion of the Investigator, might pose a risk to the subject or make participation not in the subject's best interest
* Subject is currently enrolled in or has not yet completed at least 30 days since ending another investigational device or drug study or is receiving other investigational agents
* A direct or familial relationship with the Sponsor, Investigator, or site personnel affiliated with the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (53):
- United States (44):
  - Birmingham, Alabama
  - Litchfield Park, Arizona
  - Tempe, Arizona
  - Anaheim, California
  - Chino, California
  - Chula Vista, California
  - Fresno, California
  - Gold River, California
  - Greenbrae, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Hallandale, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Avon, Indiana
  - Evansville, Indiana
  - Franklin, Indiana
  - Greenfield, Indiana
  - Council Bluffs, Iowa
  - Troy, Michigan
  - Edina, Minnesota
  - Washington, Missouri
  - Omaha, Nebraska
  - Mooresville, North Carolina
  - Morgantown, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Medford, Oregon
  - Charleston, South Carolina
  - Greer, South Carolina
  - Mt. Pleasant, South Carolina
  - Spartanburg, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - South Jordan, Utah
  - Burke, Virginia
- Canada (9):
  - Victoria, British Columbia
  - Brampton, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Mirabel, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 654 subjects were recruited at multiple sites in the United States and Canada.
Pre-assignment Details: A total of 654 subjects were screened and 297 subjects passed the run-in screening period and were randomized. One subject failed screening but was randomized in error.
Period: Overall Study
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Started | 46 | 46 | 69 | 68 | 69
Inadvertently Randomized | 0 | 0 | 0 | 1 | 0
Safety Set | 43 | 44 | 68 | 68 | 69
Modified Intent-to-Treat Set (mITT) | 40 | 38 | 61 | 62 | 62
Completed | 34 | 35 | 54 | 58 | 52
Not Completed | 12 | 11 | 15 | 10 | 17
Not completed — Adverse Event | 0 | 1 | 3 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 2 | 2 | 7
Not completed — Persistent hyperglycemia | 0 | 1 | 1 | 1 | 1
Not completed — Study terminated by sponsor | 1 | 1 | 1 | 1 | 2
Not completed — Reason not provided | 0 | 0 | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Develop anemia | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0
Not completed — Disposition Missing Due to Fire at Site | 2 | 3 | 4 | 3 | 4

BASELINE CHARACTERISTICS:
Population: All participants randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo | Total
Number analyzed (Participants) | 46 | 46 | 69 | 68 | 69 | 298
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (9.30) | 57.0 (8.95) | 57.0 (9.41) | 57.4 (7.77) | 55.6 (7.72) | 56.7 (8.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 38 | 28 | 30 | 140
  Male | 24 | 24 | 31 | 40 | 39 | 158
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 0 | 1 | 4
  Asian | 3 | 3 | 3 | 4 | 13 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 10 | 10 | 10 | 44
  White | 34 | 36 | 54 | 53 | 45 | 222
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 7 | 6 | 7 | 12 | 15 | 47
  United States | 39 | 40 | 62 | 56 | 54 | 251
1. Glycated Hemoglobin [Mean (Standard Deviation); unit: mmol/mol] — Glycated hemoglobin is a form of hemoglobin that is measured primarily to identify the three-month average glucose concentration in the blood. Target HbA1c for Type 2 diabetics was less than 7% at the time of this trial. Population: Modified Intent to Treat (mITT) Set, defined as all participants in the Safety Set who have a baseline measurement and at least 1 post-baseline measurement. mITT was used for analysis because one of the sites had a fire so 16 participants who were included in the baseline population were not included in analyses.
  mmol/mol
    number analyzed (Participants) | 40 | 38 | 61 | 62 | 62 | 263
    (all) | 7.94 (0.939) | 8.09 (0.910) | 7.99 (0.900) | 7.78 (0.790) | 7.92 (0.699) | 7.93 (0.852)
2. Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Total cholesterol is a measure of the total amount of cholesterol in the blood, including low-density lipoprotein cholesterol (LDL-C) - the "bad" cholesterol, high-density lipoprotein cholesterol (HDL-C) - the "good" cholesterol, and triglycerides. The equation to calculate total cholesterol is: LDL + HDL + (triglycerides/5) = total cholesterol. Population: Modified Intent to Treat (mITT) Set, defined as all participants in the Safety Set who have a baseline measurement and at least 1 post-baseline measurement. mITT was used for analysis because one of the sites had a fire so 16 participants who were included in the baseline population were not included in analyses.
  mg/dL
    number analyzed (Participants) | 40 | 38 | 61 | 62 | 62 | 263
    (all) | 177.1 (36.72) | 180.3 (32.21) | 178.0 (37.38) | 172.6 (55.25) | 182.8 (43.11) | 178.1 (41.70)
3. Low Density Lipoprotein-C [Mean (Standard Deviation); unit: mg/dL] — LDL-C is known as the "bad" cholesterol. Population: Modified Intent to Treat (mITT) Set, defined as all participants in the Safety Set who have a baseline measurement and at least 1 post-baseline measurement. mITT was used for analysis because one of the sites had a fire so 16 participants who were included in the baseline population were not included in analyses.
  mg/dL
    number analyzed (Participants) | 40 | 38 | 61 | 62 | 62 | 263
    (all) | 96.6 (33.58) | 96.9 (30.53) | 96.6 (32.84) | 95.1 (37.93) | 99.8 (37.14) | 97.0 (34.51)
4. High Density Lipoprotein-C [Mean (Standard Deviation); unit: mg/dL] — HDL-C is known as the "good" cholesterol. Population: Modified Intent to Treat (mITT) Set, defined as all participants in the Safety Set who have a baseline measurement and at least 1 post-baseline measurement. mITT was used for analysis because one of the sites had a fire so 16 participants who were included in the baseline population were not included in analyses.
  mg/dL
    number analyzed (Participants) | 40 | 38 | 61 | 62 | 62 | 263
    (all) | 49.5 (12.80) | 49.3 (13.20) | 46.4 (11.77) | 44.3 (12.17) | 46.7 (10.93) | 46.87 (12.19)
5. Non-High Density Lipoprotein-C [Mean (Standard Deviation); unit: mg/dL] — Non-HDL-C is the measure of "bad" cholesterol in the blood, including triglycerides and LDL-C. Population: Modified Intent to Treat (mITT) Set, defined as all participants in the Safety Set who have a baseline measurement and at least 1 post-baseline measurement. mITT was used for analysis because one of the sites had a fire so 16 participants who were included in the baseline population were not included in analyses.
  mg/dL
    number analyzed (Participants) | 40 | 38 | 61 | 62 | 62 | 263
    (all) | 127.6 (38.13) | 131.0 (32.54) | 131.6 (35.93) | 128.4 (44.46) | 136.1 (40.69) | 131.21 (38.56)
6. Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Triglycerides are a type of fat found in the blood. The body uses them for energy. Some triglycerides are needed for good health. But high triglycerides might raise the risk of heart disease. Population: Modified Intent to Treat (mITT) Set, defined as all participants in the Safety Set who have a baseline measurement and at least 1 post-baseline measurement. mITT was used for analysis because one of the sites had a fire so 16 participants who were included in the baseline population were not included in analyses.
  mg/dL
    number analyzed (Participants) | 40 | 38 | 61 | 62 | 62 | 263
    (all) | 165.3 (114.5) | 174.9 (95.55) | 179.6 (83.39) | 169.8 (84.90) | 184.2 (91.02) | 175.5 (94.54)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 12
Description: Glycated hemoglobin is a form of hemoglobin that is measured primarily to identify the three-month average glucose concentration in the blood. Target HbA1c for Type 2 diabetics was less than 7% at the time of this trial. Negative scores show improvement from baseline.
Time Frame: Baseline, Week 12
Population: Modified Intent to Treat (mITT) Set, defined as all participants in the Safety Set who have a baseline measurement and at least 1 post-baseline measurement. mITT was used for analysis because one of the sites had a fire so 16 participants who were included in the baseline population were not included in analyses.
Measure: Mean (Standard Deviation); unit: percent of HbA1c
Groups:
- DS-8500a 25mg: One DS-8500a 25 mg tablets and placebo
- DS-8500a 50 mg: Two DS-8500a 25 mg tablets and placebo
- DS-8500a 75 mg: Three DS-8500a 25 mg tablets and placebo
- Sitagliptin 100 mg: One sitagliptin 100 mg over-capsule and placebo
- Placebo: Placebo tablets and capsule
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 35 | 33 | 53 | 57 | 53
percent of HbA1c | -0.24 (1.019) | -0.16 (0.798) | -0.35 (0.791) | -0.66 (0.623) | -0.23 (0.657)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 12; Test type: Other; p = .755, Mixed Model Repeated Measure; LS Mean Difference = 0.05, 90% CI 2-sided [-0.211 to 0.309], Standard Error of Mean 0.157
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .512, Mixed Model Repeated Measure; LS Mean Difference = 0.11, 90% CI 2-sided [-0.160 to 0.371], Standard Error of Mean 0.161
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .566, Mixed Model Repeated Measure; LS Mean Difference = -0.08, 90% CI 2-sided [-0.312 to 0.151], Standard Error of Mean 0.140
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .002, Mixed Model Repeated Measure; LS Mean Difference = -0.43, 90% CI 2-sided [-0.655 to -0.197], Standard Error of Mean 0.139

2. Secondary Outcome: Change From Baseline in Total Cholesterol (TC) at Week 12
Description: Total cholesterol is a measure of the total amount of cholesterol in the blood, including low-density lipoprotein cholesterol (LDL-C) - the "bad" cholesterol, high-density lipoprotein cholesterol (HDL-C) - the "good" cholesterol, and triglycerides. The equation to calculate total cholesterol is: LDL + HDL + (triglycerides/5) = total cholesterol.
Time Frame: Baseline, Week 12
Population: mITT
Measure: Mean (Standard Deviation); unit: percent change in TC
Groups:
- DS-8500a 25mg: One DS-8500a 25 mg tablet and placebo
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 34 | 33 | 52 | 57 | 51
percent change in TC | -5.6 (11.95) | -1.7 (22.30) | -1.8 (12.58) | -3.6 (14.34) | -1.7 (13.57)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 12; Test type: Other; p = .144, Mixed Model Repeated Measure; LS Mean Difference = -4.6, 90% CI 2-sided [-9.76 to 0.58], Standard Error of Mean 3.13
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .773, Mixed Model Repeated Measure; LS Mean Difference = -0.9, 90% CI 2-sided [-6.14 to 4.31], Standard Error of Mean 3.16
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .963, Mixed Model Repeated Measure; LS Mean Difference = -0.1, 90% CI 2-sided [-4.73 to 4.48], Standard Error of Mean 2.79
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .258, Mixed Model Repeated Measure; LS Mean Difference = -3.1, 90% CI 2-sided [-7.64 to 1.42], Standard Error of Mean 2.74

3. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Description: LDL-C is known as the "bad" cholesterol, so a lower score (negative change) means improvement.
Time Frame: Baseline, Week 12
Population: mITT
Measure: Mean (Standard Deviation); unit: percent change in LDL-C
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 33 | 33 | 52 | 57 | 50
percent change in LDL-C | -6.7 (17.34) | 2.8 (46.18) | -0.1 (22.84) | -2.4 (23.20) | 0.9 (20.12)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 12; Test type: Other; p = .228, Mixed Model Repeated Measure; LS Mean Difference = -6.7, 90% CI 2-sided [-15.74 to 2.43], Standard Error of Mean 5.50
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .894, Mixed Model Repeated Measure; LS Mean Difference = 0.7, 90% CI 2-sided [-8.36 to 9.84], Standard Error of Mean 5.51
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .846, Mixed Model Repeated Measure; LS Mean Difference = -0.9, 90% CI 2-sided [-8.97 to 7.08], Standard Error of Mean 4.86
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .409, Mixed Model Repeated Measure; LS Mean Difference = -3.9, 90% CI 2-sided [-11.82 to 3.93], Standard Error of Mean 4.77

4. Secondary Outcome: Change From Baseline in HDL-C at Week 12
Description: HDL-C is known as the "good" cholesterol, so a higher score (positive change) means improvement.
Time Frame: Baseline, Week 12
Population: mITT
Measure: Mean (Standard Deviation); unit: percent change in HCL-C
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 34 | 33 | 52 | 57 | 51
percent change in HCL-C | 3.0 (11.48) | 1.1 (10.18) | 2.2 (11.59) | 1.1 (13.17) | 1.2 (11.41)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 12; Test type: Other; p = .576, Mixed Model Repeated Measure; LS Mean Difference = 1.5, 90% CI 2-sided [-2.83 to 5.73], Standard Error of Mean 2.59
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .646, Mixed Model Repeated Measure; LS Mean Difference = -1.2, 90% CI 2-sided [-5.53 to 3.12], Standard Error of Mean 2.62
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .902, Mixed Model Repeated Measure; LS Mean Difference = 0.3, 90% CI 2-sided [-3.52 to 4.08], Standard Error of Mean 2.30
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .478, Mixed Model Repeated Measure; LS Mean Difference = -1.6, 90% CI 2-sided [-5.35 to 2.13], Standard Error of Mean 2.27

5. Secondary Outcome: Change From Baseline in Non-HDL-C at Week 12
Description: Non-HDL-C is the measure of "bad" cholesterol in the blood, including triglycerides and LDL-C, so a negative change means improvement. The equation for Non-HDL-C = LDL-C + (triglycerides/5).
Time Frame: Baseline, Week 12
Population: mITT
Measure: Mean (Standard Deviation); unit: Percent change in Non-HDL-C
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 34 | 33 | 52 | 57 | 51
Percent change in Non-HDL-C | -8.9 (14.89) | -2.5 (31.68) | -2.9 (16.68) | -4.7 (19.10) | -2.5 (17.02)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 12; Test type: Other; p = .072, Mixed Model Repeated Measure; LS Mean Difference = -7.6, 90% CI 2-sided [-14.57 to -0.64], Standard Error of Mean 4.22
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .794, Mixed Model Repeated Measure; LS Mean Difference = -1.1, 90% CI 2-sided [-8.15 to 5.92], Standard Error of Mean 4.26
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .946, Mixed Model Repeated Measure; LS Mean Difference = -0.3, 90% CI 2-sided [-6.45 to 5.94], Standard Error of Mean 3.75
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .431, Mixed Model Repeated Measure; LS Mean Difference = -2.9, 90% CI 2-sided [-8.99 to 3.18], Standard Error of Mean 3.68

6. Secondary Outcome: Change From Baseline in Triglycerides at Week 12
Description: Triglycerides are a type of fat found in the blood. The body uses them for energy. Some triglycerides are needed for good health. But high triglycerides might raise the risk of heart disease. Since Type 2 diabetics tend to have high triglycerides, a negative change means improvement.
Time Frame: Baseline, Week 12
Population: mITT
Measure: Mean (Standard Deviation); unit: percent change in triglycerides
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 34 | 33 | 52 | 57 | 51
percent change in triglycerides | -12.4 (22.35) | -1.9 (78.27) | -5.8 (27.71) | -7.0 (27.90) | -3.0 (27.76)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 12; Test type: Other; p = .228, Mixed Model Repeated Measure; LS Mean Difference = -10.3, 90% CI 2-sided [-24.43 to 3.78], Standard Error of Mean 8.54
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .951, Mixed Model Repeated Measure; LS Mean Difference = 0.5, 90% CI 2-sided [-13.70 to 14.77], Standard Error of Mean 8.62
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .852, Mixed Model Repeated Measure; LS Mean Difference = -1.4, 90% CI 2-sided [-13.96 to 11.13], Standard Error of Mean 7.59
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .608, Mixed Model Repeated Measure; LS Mean Difference = -3.8, 90% CI 2-sided [-16.13 to 8.48], Standard Error of Mean 7.45

7. Secondary Outcome: Change From Baseline in Area-Under-the Curve 0-3 Hours (AUC0-3h) of Plasma Glucose (PG) in Response to the Mixed Meal Tolerance Test (MMTT) at Week 4
Description: The MMTT requires a participant to drink a "mixed meal," such as Boost or Ensure, that contains protein, carbohydrates, and fat. The goal of the test is to find out how much insulin the pancreas makes in response to food by measuring the level of glucose in the blood. The lower the level of glucose in the blood during the first three hours after the test (AUC0-3h), the more insulin the body has made in response to the test. This would mean a negative change shows improvement.
Time Frame: Baseline, Week 4
Population: mITT with a measurement at baseline and Week 4
Measure: Mean (Standard Deviation); unit: (mg/dL)*hr
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 37 | 35 | 55 | 59 | 57
(mg/dL)*hr | -4.32 (71.235) | 1.36 (67.661) | -6.32 (83.597) | -41.61 (73.971) | -3.97 (87.625)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 4; Test type: Other; p = .728, Mixed Model Repeated Measure; LS Mean Difference = 5.32, 90% CI 2-sided [-19.932 to 30.566], Standard Error of Mean 15.289
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 4; Test type: Other; p = .837, Mixed Model Repeated Measure; LS Mean Difference = -3.27, 90% CI 2-sided [-29.446 to 22.914], Standard Error of Mean 15.853
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 4; Test type: Other; p = .791, Mixed Model Repeated Measure; LS Mean Difference = -3.65, 90% CI 2-sided [-26.352 to 19.051], Standard Error of Mean 13.747
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 4; Test type: Other; p = .003, Mixed Model Repeated Measure; LS Mean Difference = -40.03, 90% CI 2-sided [-62.283 to -17.787], Standard Error of Mean 13.472

8. Secondary Outcome: Change From Baseline in AUC0-3h of PG in Response to the MMTT at Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 12
Population: mITT with a measurement at baseline and Week 12
Measure: Mean (Standard Deviation); unit: (mg/dL)*hr
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 28 | 31 | 47 | 51 | 49
(mg/dL)*hr | -18.77 (96.472) | 13.81 (67.025) | -5.51 (104.992) | -53.40 (74.803) | -24.16 (101.016)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 12; Test type: Other; p = .830, Mixed Model Repeated Measure; LS Mean Difference = 4.39, 90% CI 2-sided [-29.312 to 38.087], Standard Error of Mean 20.396
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .235, Mixed Model Repeated Measure; LS Mean Difference = 24.25, 90% CI 2-sided [-9.354 to 57.848], Standard Error of Mean 20.335
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .331, Mixed Model Repeated Measure; LS Mean Difference = 17.25, 90% CI 2-sided [-12.030 to 46.529], Standard Error of Mean 17.720
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .091, Mixed Model Repeated Measure; LS Mean Difference = -29.51, 90% CI 2-sided [-58.254 to -0.775], Standard Error of Mean 17.393

9. Secondary Outcome: Change From Baseline in Maximum Concentration (Cmax) of PG in Response to MMTT at Week 4
Description: Cmax measures the highest amount of glucose in the blood, so a negative change means improvement.
Time Frame: Baseline, Week 4
Population: mITT with a measurement at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 37 | 35 | 56 | 59 | 57
mg/dL | -1.92 (41.260) | -7.35 (39.645) | -3.47 (54.258) | -28.44 (45.327) | -0.35 (41.885)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 4; Test type: Other; p = .873, Mixed Model Repeated Measure; LS Mean Difference = 1.49, 90% CI 2-sided [-13.835 to 16.815], Standard Error of Mean 9.280
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 4; Test type: Other; p = .395, Mixed Model Repeated Measure; LS Mean Difference = -8.09, 90% CI 2-sided [-23.790 to 7.604], Standard Error of Mean 9.505
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 4; Test type: Other; p = .761, Mixed Model Repeated Measure; LS Mean Difference = -2.53, 90% CI 2-sided [-16.247 to 11.185], Standard Error of Mean 8.306
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 4; Test type: Other; p < 0.001, Mixed Model Repeated Measure; LS Mean Difference = -27.73, 90% CI 2-sided [-41.220 to -14.236], Standard Error of Mean 8.170

10. Secondary Outcome: Change From Baseline in Cmax of PG in Response to MMTT at Week 12
Description: Cmax measures the highest amount of glucose in the blood, so a negative change means improvement.
Time Frame: Baseline, Week 12
Population: mITT with a measurement at baseline and Week 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 28 | 31 | 47 | 51 | 49
mg/dL | -5.93 (47.530) | -1.10 (53.045) | -4.43 (60.957) | -28.29 (42.184) | 1.11 (58.731)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 12; Test type: Other; p = .527, Mixed Model Repeated Measure; LS Mean Difference = -7.61, 90% CI 2-sided [-27.441 to 12.221], Standard Error of Mean 12.001
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .532, Mixed Model Repeated Measure; LS Mean Difference = -7.39, 90% CI 2-sided [-26.927 to 12.138], Standard Error of Mean .532
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .672, Mixed Model Repeated Measure; LS Mean Difference = -4.41, 90% CI 2-sided [-21.635 to 12.807], Standard Error of Mean 10.421
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .002, Mixed Model Repeated Measure; LS Mean Difference = -31.58, 90% CI 2-sided [-48.482 to -14.676], Standard Error of Mean 10.229

11. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 2
Description: Normal fasting plasma glucose -- or blood sugar -- is between 70 and 100 milligrams per deciliter (mg/dL) for people who do not have diabetes. People with Type 2 diabetes typically have FPG that is too high, so a negative change from baseline means improvement.
Time Frame: Baseline, Week 2
Population: mITT with a measurement at baseline and Week 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 40 | 36 | 58 | 57 | 58
mg/dL | 4.3 (25.98) | -8.1 (25.24) | 0.0 (31.52) | -16.2 (26.11) | 10.7 (32.38)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 2; Test type: Other; p = .298, Mixed Model Repeated Measure; LS Mean Difference = -6.2, 90% CI 2-sided [-15.90 to 3.60], Standard Error of Mean 5.90
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 2; Test type: Other; p = .008, Mixed Model Repeated Measure; LS Mean Difference = -16.3, 90% CI 2-sided [-26.37 to -6.27], Standard Error of Mean 6.09
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 2; Test type: Other; p = .074, Mixed Model Repeated Measure; LS Mean Difference = -9.5, 90% CI 2-sided [-18.31 to -0.75], Standard Error of Mean 5.32
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 2; Test type: Other; p < 0.001, Mixed Model Repeated Measure; LS Mean Difference = -27.2, 90% CI 2-sided [-35.96 to -18.38], Standard Error of Mean 5.32

12. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 4
Description: as for outcome 11
Time Frame: Baseline, Week 4
Population: mITT with a measurement at baseline and Week 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 60 | 62 | 62
mg/dL | 0.04 (18.71) | -12.7 (30.82) | -5.9 (35.17) | -11.1 (31.81) | 2.4 (32.01)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 4; Test type: Other; p = .840, Mixed Model Repeated Measure; LS Mean Difference = -1.2, 90% CI 2-sided [-11.04 to 8.63], Standard Error of Mean 5.96
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 4; Test type: Other; p = .050, Mixed Model Repeated Measure; LS Mean Difference = -11.9, 90% CI 2-sided [-21.94 to -1.91], Standard Error of Mean 6.06
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 4; Test type: Other; p = .227, Mixed Model Repeated Measure; LS Mean Difference = -6.4, 90% CI 2-sided [-15.21 to 2.33], Standard Error of Mean 5.31
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 4; Test type: Other; p = 0.13, Mixed Model Repeated Measure; LS Mean Difference = -13.1, 90% CI 2-sided [-21.83 to -4.43], Standard Error of Mean 5.27

13. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 8
Description: as for outcome 11
Time Frame: Baseline, Week 8
Population: mITT with a measurement at baseline and Week 8
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 36 | 33 | 56 | 56 | 55
mg/dL | 2.3 (27.57) | -5.9 (27.90) | -7.1 (37.51) | -16.6 (32.96) | -1.0 (31.63)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 8; Test type: Other; p = .642, Mixed Model Repeated Measure; LS Mean Difference = 3.1, 90% CI 2-sided [-7.77 to 13.88], Standard Error of Mean 6.55
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 8; Test type: Other; p = .512, Mixed Model Repeated Measure; LS Mean Difference = -4.4, 90% CI 2-sided [-15.52 to 6.68], Standard Error of Mean 6.72
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 8; Test type: Other; p = .486, Mixed Model Repeated Measure; LS Mean Difference = -4.1, 90% CI 2-sided [-13.66 to 5.54], Standard Error of Mean 5.81
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 8; Test type: Other; p = .004, Mixed Model Repeated Measure; LS Mean Difference = -16.7, 90% CI 2-sided [-26.31 to -7.16], Standard Error of Mean 5.80

14. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12
Description: as for outcome 11
Time Frame: Baseline, Week 12
Population: mITT with a measurement at baseline and Week 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 28 | 31 | 47 | 52 | 49
mg/dL | 0.0 (25.67) | -9.1 (34.89) | -5.8 (35.27) | -5.7 (46.29) | 8.1 (32.72)
Statistical Analysis 1: Comparison: DS-8500a 25mg vs Placebo; Difference in change at week 12; Test type: Other; p = .285, Mixed Model Repeated Measure; LS Mean Difference = -8.7, 90% CI 2-sided [-22.09 to 4.70], Standard Error of Mean 8.11
Statistical Analysis 2: Comparison: DS-8500a 50 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .020, Mixed Model Repeated Measure; LS Mean Difference = -18.6, 90% CI 2-sided [-31.73 to -5.49], Standard Error of Mean 7.94
Statistical Analysis 3: Comparison: DS-8500a 75 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .067, Mixed Model Repeated Measure; LS Mean Difference = -13.0, 90% CI 2-sided [-24.60 to -1.35], Standard Error of Mean 7.03
Statistical Analysis 4: Comparison: Sitagliptin 100 mg vs Placebo; Difference in change at week 12; Test type: Other; p = .012, Mixed Model Repeated Measure; LS Mean Difference = -17.4, 90% CI 2-sided [-28.76 to -6.03], Standard Error of Mean 6.88

15. Secondary Outcome: Count of Participants With HbA1c Less Than 7.0% at Week 12
Description: HbA1C less than 7% is the success goal for many Type 2 diabetics.
Time Frame: Week 12
Population: mITT
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo tablets and placebo capsule
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 40 | 38 | 61 | 62 | 62
Participants | 6 | 8 | 15 | 28 | 10

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that first occurred or worsened in severity after initiation of double-blind treatment, were collected until the end of treatment (12 weeks), plus two weeks of follow-up.
Arm/Group | DS-8500a 25mg | DS-8500a 50 mg | DS-8500a 75 mg | Sitagliptin 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44 | 0/68 | 0/68 | 0/69
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/44 | 1/68 | 1/68 | 0/69
Other Adverse Events (participants affected / at risk) | 7/43 | 2/44 | 11/68 | 6/68 | 7/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DS-8500a 25mg (N=43) | DS-8500a 50 mg (N=44) | DS-8500a 75 mg (N=68) | Sitagliptin 100 mg (N=68) | Placebo (N=69)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DS-8500a 25mg (N=43) | DS-8500a 50 mg (N=44) | DS-8500a 75 mg (N=68) | Sitagliptin 100 mg (N=68) | Placebo (N=69)
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 4 | 3 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 4
Nausea (Gastrointestinal disorders) | 3 | 0 | 4 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 2 | 2 | 1

LIMITATIONS AND CAVEATS:
Accidental fire at one site changed the baseline number of participants for the modified intent to treat (mITT) set. Because of this, baseline data were included in the outcome measures, rather than in the baseline module.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT02647320/Prot_SAP_000.pdf